CLINICAL TRIAL: NCT04291989
Title: Optimal Blood Sampling Site for Point of Care Lactate Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Edge I.D - 90666
Record Dates: First submitted 2020-02-26; First posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Blood Lactic Acid Increased; Hip Fractures
Keywords: BLOOD LACTATE; EARLOBE SAMPLE; FINGER PRICK SAMPLE
MeSH Terms: conditions — Hyperlactatemia; Hip Fractures

STUDY DESIGN:
Intervention Model Description: This study aims to compare lactate levels from the same patient at the same time with blood samples taken from three locations - fingertip, earlobe and forearm venepuncture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Earlobe and Finger Prick versus venous blood lactate sampling (Experimental): Compare blood Lactate levels between ear lobe and finger against venous forearm blood sample using the electronic hand held lactate device in hip fracture patients with good cognitive function (AMT >/= 7)
  Interventions: Device: Optimal Blood Sampling Site for Point of Care Lactate Assessment using the handled Lactate-Pro 2 device

INTERVENTIONS:
Device: Optimal Blood Sampling Site for Point of Care Lactate Assessment using the handled Lactate-Pro 2 device — This study aims to compare lactate levels using the Lactate Pro 2 device from the same patient at the same time with blood samples taken from three locations - fingertip, earlobe and forearm venepuncture

SUMMARY:
The study was to compare blood Lactate levels between ear lobe and finger against venous forearm blood sample using the electronic hand held lactate device in hip fracture patients with good cognitive function (AMT >/= 7)

DETAILED DESCRIPTION:
Following a hip fracture, surgical treatment is advocated to improve pain and mobility. Most patients are elderly and a majority of them are frail. Current best practice tariff and National Institute for health and care excellence guidelines recommends that all those patients who undergo an operation should be performed within 36 hours from the time of injury to optimise recovery and function. The patients need to be medically optimised to undergo a major operation to have their hip fracture fixed. The adequacy of resuscitation is monitored by several clinical and biochemical markers. One of the important markers of resuscitation is serum lactate levels. This is used routinely in polytrauma patients. (Moran and Forward, 2012) The initial interest in lactate in hip fracture patients was based on the philosophy that a hip fracture in a frail elderly patient may be equivalent to a polytrauma in a young fit patient. Subsequently, high serum lactate levels on admission in hip fracture patients have been shown to be associated with higher mortality1. However, at present, this is not routinely monitored in hip fracture patients. Measurement of serum lactate levels presents logistics difficulties, as the blood sample has to be taken to an analyser and analysed within 20 minutes. Hence the investigators want to use a point of care electronic hand held device - the Lactate Pro 2. The investigators have already tested this device against the laboratory analysers and it has been proven to be accurate. However in preliminary testing the investigators found a significant difference between fingertip and earlobe samples in volunteers. The volunteers do not represent our population of interest, which are hip fracture patients. The investigators aim is to determine which sample site; earlobe or fingertip, for Lactate Pro 2 testing best matches venous forearm samples upon which the association of higher mortality with high lactate was based.

Any risk to the patients participating in this study would be very small. The inclusion criteria to participate in this research study is a patient who has had a recent hip fracture awaiting surgery with a Mental Test score of 7/10 or above and is able to consent.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged 18 years or above.
* Diagnosed with an acute hip fracture.
* Have a mental test score of 7/10 or greater on assessment during admission.
* Participant is willing to consent to the study.

Exclusion Criteria:

* The participant will not enter the study if

  1. There are Injuries other than isolated hip fracture
  2. Age <18 years
  3. They are not willing to consent for the study
  4. They have a mental test score less than 7/10 at the time of admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Finger prick blood sample and earlobe prick blood sample compared to forearm venepuncture blood sample to measure blood Lactate levels in mmol/l using the point of care Lactate-Pro2 device | The investigators aim to recruit 50 acute hip fracture patients over a time period of upto 6 months for our study. The outcome will be measured only once and recorded at the point of care for each patient.
  Which of the two sample sites - finger or earlobe most closely matches the forearm venepuncture blood sample for measuring blood lactate levels?

CONTACTS AND LOCATIONS:
Overall Officials: GANAPATHY RAMAN R Perianayagam, FRCS (Orth), Principal Investigator — University Hospitals, Leicester
Locations (1):
- Leicester Royal Infirmary, Leicester, Please Select, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant date for primary outcomes will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: for 6 months after publication of the study
Access Criteria: Data access will be reviewed by an external review panel. Requestors will be required to sign a Data Access Agreement form.